CLINICAL TRIAL: NCT03947138
Title: A Multi-national, Multi-center, Randomized, Double-Blind, Active-Controlled, Phase III Study to Investigate the Efficacy and Safety of 'GC3107(BCG Vaccine)' After Intradermal Administration in Healthy Infants
Brief Title: A Study of GC3107(BCG Vaccine) in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3107_P3
Record Dates: First submitted 2019-04-29; First posted 2019-05-13 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: BCG Vaccination Reaction; Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GC3107_Part1 (Experimental): Part 1 GC3107(BCG Vaccine) Single intradermal Injection of 0.05 mL into the end of deltoid muscle in outer aspect of upper arm
  Interventions: Biological: GC3107
- GC3107_Part2 (Experimental): Part 2 GC3107(BCG Vaccine) Single intradermal Injection of 0.05 mL into the end of deltoid muscle in outer aspect of upper arm
  Interventions: Biological: GC3107
- BCG SSI_Part1 (Active Comparator): Part 1 Intradermal BCG SSI inj Single intradermal Injection of 0.05 mL into the end of deltoid muscle in outer aspect of upper arm
  Interventions: Biological: Intradermal BCG SSI inj.
- BCG SSI_Part2 (Active Comparator): Part 2 Intradermal BCG SSI inj Single intradermal Injection of 0.05 mL into the end of deltoid muscle in outer aspect of upper arm
  Interventions: Biological: Intradermal BCG SSI inj.

INTERVENTIONS:
Biological: GC3107 — BCG Vaccine
  Arms: GC3107_Part1; GC3107_Part2
Biological: Intradermal BCG SSI inj. — BCG Vaccine
  Arms: BCG SSI_Part1; BCG SSI_Part2

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of GC3107 in healthy infants

DETAILED DESCRIPTION:
The study will be conducted in 2 Countries, Korea and Thailand. About 750 subjects will be enrolled to this study.

This clinical trial consists of Part 1 to compare the efficacy and safety between the study group and the active control group and Part 2 for the final safety assessment. Subject enrollment for Part 1 and Part 2 will occur at the same time, and subjects who meet the final inclusion/exclusion criteria will be randomized to Part 1 or Part 2 via the IWRS.

When the legally acceptable representative of the subject within 4 weeks after birth consents to participate in the clinical study in writing at Visit 1, the protocol-mandated examination and tests will be performed at each visit, and only the subjects who meet the inclusion/exclusion criteria will be assigned randomization numbers and receive a single intradermal injection of the investigational product. However, the informed consent of the subject's legally acceptable representative for participation in the clinical trial may be obtained between 36 weeks of pregnancy of a subject's mother and Visit 1.

The investigator will instruct the subject's legally acceptable representative to record any adverse events (AEs) occurring after administration of the investigational product to assess the safety of the subject during the study period.

The subjects participating in Part 1 will have the tuberculin skin test at Visit 4 for the efficacy assessment and receive an intradermal injection of 0.1 mL purified protein derivatives (PPD) reagent. Visit 5 will occur within 48 to 72 hours of the PPD reagent injection to check the tuberculin skin test results.

Also, Visit 6 will be conducted as an on-site visit to check for any solicited local AEs (abscess, ulcer, scar, and BCG lymphadenitis) and unsolicited AEs occurring until 6 months (168 days) after administration of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's legally acceptable representatives had this clinical trial information explained to them and understood it, voluntarily decided participation, and provided informed consent
2. Healthy infants aged≤4weeks
3. Body weight≥2,500g at birth
4. Born after normal gestation(≥37weeks)

Exclusion Criteria:

1. Had contact with patients with a confirmed diagnosis of active pulmonary tuberculosis
2. Any symptoms or signs of active tuberculosis infection or current treatment of tuberculosis at screening
3. History of confirmed tuberculosis
4. Acute fever with tympanic temperature≥38.0 'C within 24 hours prior to administration of the investigational product, or an active infections disease at screening
5. Hypothermia with tympanic temperature<36.0 'C within 24 hours prior to administration of the investigational product
6. Clinically suspected neonatal sepsis
7. Born with severe congenital anomaly that may affect the efficacy or safety result of this clinical trial as judged by the investigator
8. Severe skin disease or burn at the injection site of investigational product
9. The subject's mother had human immunodeficiency virus (HIV)-positive result on prenatal testing

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-09-06 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with maximum diameter of induration ≥ 5mm in the tuberculin skin test | 84 days after administration of the investigational product
  Induration diameter measured in the direction perpendicular to the arm.

SECONDARY OUTCOMES:
Proportion of subjects with maximum diameter of induration <5mm, ≥ 5mm to <10mm and ≥10mm in the tuberculin skin test | 84 days after administration of the investigational product
  Induration diameter measured in the direction perpendicular to the arm.
Proportion of subjects with maximum diameter of erythema ≥ 5mm in the tuberculin skin test | 84 days after administration of the investigational product
  Erythema diameter measured in the direction perpendicular to the arm.

CONTACTS AND LOCATIONS:
Overall Officials: JongHyun Kim, MD, Principal Investigator — The Catholic University of Korea St. Vincent's Hospital, Pediatrics
Locations (2):
- South Korea (2):
  - The Catholic Universitiy of Korea St. vincent's Hospital, Suwon
  - Greencross, Yŏngin